CLINICAL TRIAL: NCT04932291
Title: "A Double-blind, Randomized, Placebo-controlled, Adaptive 14-week Phase IIb Trial to Evaluate the Efficacy and Safety of Vafidemstat in an Adult Borderline Personality Disorder (BPD) Population (PORTICO)"
Brief Title: Study to Test the Efficacy and Safety of Vafidemstat in Adult Borderline Personality Disorder Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oryzon Genomics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL07-ORY-2001
Record Dates: First submitted 2021-04-12; First posted 2021-06-21 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-09

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline personality disorder; vafidemstat
MeSH Terms: conditions — Borderline Personality Disorder | interventions — vafidemstat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- vafidemstat 1.2mg (Experimental): Vafidemstat is administered as capsules.
  Interventions: Drug: vafidemstat
- placebo (Placebo Comparator): Placebo is administered as capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vafidemstat — 1.2mg capsule
  Other Names: ORY-2001
  Arms: vafidemstat 1.2mg
Drug: Placebo — placebo capsule
  Arms: placebo

SUMMARY:
PORTICO is a Phase IIb study to evaluate the efficacy and safety of vafidemstat in an adult borderline personality disorder (BPD) population.

DETAILED DESCRIPTION:
PORTICO is a double blind, randomized, placebo-controlled, adaptive 14-week Phase IIb trial to evaluate the efficacy and safety of vafidemstat in an adult borderline personality disorder (BPD) population.

ELIGIBILITY:
Principal inclusion criteria:

1. Men and women 18-65 years of age.
2. DSM-5 diagnostic criteria for BPD at least 3 months before the Screening visit. The Mini-International Neuropsychiatric Interview (MINI) will be administered at screening in order to confirm BPD diagnosis, as well as to confirm subject does not meet other relevant exclusion criteria.
3. Agitation-Aggression Psychiatric Inventory-Clinician Report (AAPI-CR) Agitation & Aggression (A/A) subscale score of > 16 (severity x frequency) summed across the four (4) items comprising the A/A subscale, and the sum of the A/A subscale severity scores > 6.
4. Outpatient known to the site or investigator and has been treated by the site or investigator for at least the last 3 months prior to the Screening visit.
5. Stable living environment for > 6 months before the Screening visit.
6. Body mass index (BMI) of at least 18.5 kg/m2, but no more than 35 kg/m2.
7. Willing and able to adhere to the prohibitions, restrictions and requirements specified in this protocol.
8. Otherwise, healthy, and medically stable based on medical history.
9. Clinical and neurological examinations and laboratory tests, as well as 12-lead ECG performed during screening that confirms subject is healthy and medically stable.
10. Able to read and write fluently and must have adequate hearing and visual acuity to complete the required testing outlined in this protocol.
11. Stable in their permitted regimen of background therapy as per drug labeling for concomitant medications at the Screening visit and they should maintain treatment throughout the study and not initiate any prohibited medications during the trial. Subjects should agree to inform their study physician of any medication changes throughout the trial.
12. Enrolled subjects will need to maintain their pre-screening psychotherapy schedule throughout the trial duration. That is, subjects receiving psychotherapy will need to have it started at least 3 months before the Screening visit and remain in psychotherapy throughout the trial. Subjects not receiving psychotherapy should not initiate psychotherapy during the trial.
13. Fertile male and female subjects must use highly efficient contraception, from the Screening visit until 30 days after last dose of the IMP, defined as:

    A method with less than 1% failure rate (e.g., permanent sterilization, hormone implants, hormone injections, some intrauterine devices, or vasectomized partner) OR The use of two methods of contraception (e.g., one barrier method [condom, diaphragm or cervical/vault caps] with spermicide and one hormonal contraceptive [e.g., combined oral contraceptives, patch, vaginal ring, injectable and implants])
14. Female subjects of childbearing potential must have a negative urine pregnancy test at screening and baseline.
15. Signed informed consent by participant prior to the initiation of any study specific procedure.

Principal exclusion criteria

1. DSM-5 diagnosis of intellectual disability, autism spectrum disorder, schizophrenia, schizoaffective disorder, bipolar disorder (or related disorders) or major depressive disorder (MDD) with psychosis.
2. Current DSM-5 diagnosis of conduct disorder, anorexia nervosa, bulimia nervosa, binge-eating disorder, oppositional defiant disorder, paranoid personality disorder or obsessive-compulsive disorder.
3. Current DSM-5 diagnosis of panic disorder or post-traumatic stress disorder (PTSD). However, subjects with PTSD, generalized anxiety disorder (GAD), social anxiety disorder (SAD), MDD without psychosis, attention deficit hyperactivity disorder (ADHD) are eligible if symptoms have been stable for at least 90 days prior to the Screening visit, these disorders are not the primary focus of treatment, changes in any treatment for these disorders would not likely be required for the duration of the study, and in the investigator´s opinion these disorders will not interfere with the assessment and/or accuracy of the study endpoints.
4. History of moderate or severe substance or alcohol use disorder according to DSM-5, with the exception of nicotine and caffeine, within 6-months before screening.
5. Use of illicit drugs for at least one week before Screening and subjects unwilling to abstain from use of these substances during the study.
6. Hospitalization or medication change for any reason, two months prior to the Screening visit or during the Screening period, that makes the subject medically or mentally unsuitable for trial participation.
7. Clinically significant, advanced or unstable disease that is likely to result in rapid deterioration of the subject's condition or affect their safety during the study.
8. Positive results for tuberculosis, Human Immunodeficiency Virus (HIV), Hepatitis C or Hepatitis B serology obtained at the Screening Visit.
9. Uncontrolled hypo- or hyperthyroidism at Screening Visit, based on laboratory parameters.
10. Clinically significant infection within the previous 30-days.
11. Chronic drug intake of specific forbidden medication
12. Esketamine in the past 90 days before the Screening visit.
13. Electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) in the past 90 days before the screening visit.
14. Any regular intake of medications acting directly on central nervous system that investigator considers relevant to the study.
15. Member or immediate family of the study personnel or subordinate to any of the study personnel.
16. Enrollment in another investigational study or intake of investigational drug within the previous 3 months.
17. Suicide attempt within the 6-month prior to the Screening visit or significant risk of suicide.
18. Any condition that in the opinion of the investigator makes the subject unsuitable for inclusion in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Efficacy: Clinical Global Impression-Severity focused on Agitation/Aggression (CGI-S A/A) | From baseline up to week 14
  Evaluation of the difference on the Clinical Global Impression-Severity focused on Agitation/Aggression (CGI-S A/A) from baseline to specific week, between the active treatment arm and the placebo arm
Efficacy: Borderline Personality Disorder Checklist (BPDCL) | From baseline up to week 14
  Evaluation of the difference on the Borderline Personality Disorder Checklist (BPDCL), from baseline to specific week, between the active treatment arm and the placebo arm

SECONDARY OUTCOMES:
Efficacy: Clinical Global Impression-Severity focused on Agitation/Aggression (CGI-S A/A) | Change up to week 14
  Evaluation of the change over time on the CGI-S A/A
Efficacy: Borderline Personality Disorder Checklist (BPDCL) | Change up to week 14
  Evaluation of the change over time on the BPDCL
Efficacy: Borderline Evaluation of Severity over Time (BEST) | Change up to week 14 and from baseline to week 14
  Evaluation of the difference on BEST between the active treatment arm and the placebo arm
Efficacy: Beck Depression Inventory II (BDI-II) | Change up to week 14 and from baseline to week 14
  Evaluation of the difference on BDI-II between the active treatment arm and the placebo arm
Efficacy: State-Trait Anger Expression Inventory 2 (STAXI-2) | Change up to week 14 and from baseline to week 14
  Evaluation of the difference on STAXI-2 between the active treatment arm and the placebo arm
Efficacy: State-Trait Anxiety Inventory (STAI) | Change up to week 14 and from baseline to week 14
  Evaluation of the difference on STAI between the active treatment arm and the placebo arm
Safety - Adverse events | From baseline to week 14
  Treatment emergent adverse events
Safety - Withdrawn patients | From baseline to week 14
  Percentage of withdrawn patients
Safety endpoints - Columbia-Suicide Severity Rating Scale (C-SSRS). | From baseline to week 14
  Columbia-Suicide Severity Rating Scale (C-SSRS)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ropacki, MD, Study Director — Oryzon Genomics
Locations (21):
- United States (11):
  - Excell Research Inc, Oceanside, California
  - Excell Research, Inc., Oceanside, California
  - New Life Medical Research Center, Hialeah, Florida
  - Phoenix Medical Research LLC, Miami, Florida
  - University of Chicago Institutional Review Board, Chicago, Illinois
  - Revive Research Institute, Elgin, Illinois
  - Adams Clinical Trials, LLC, Watertown, Massachusetts
  - Center for Emotioal Fitness, Cherry Hill, New Jersey
  - Neurobehavioral Research Inc., Cedarhurst, New York
  - The Medical Research Network, New York, New York
  - Core Clinical Research, Everett, Washington
- Bulgaria (3):
  - Medical Center Intermedika, Sofia, Sofia-Grad
  - Medical Center Hera EOOD - Psychiatry Office, Sofia, Sofia-Grad
  - DCC "Mladost-M" Ltd, Psychiatr, Varna
- Germany (2):
  - Klinik fur Psychiatrie und Psychotherapie, LMU, München, Bavaria
  - Emovis GmbH, Berlin
- Serbia (3):
  - Clinic for psychiatric disorders "Laza Lazarevic", Belgrade
  - Clinical center of Serbia, Belgrade
  - Clinical center Kragujevac, Kragujevac
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No